CLINICAL TRIAL: NCT00222391
Title: Influence of Thoracic Epidural Anesthesia on Skin Sympathetic Activity and Heart Rate Variability in Surgical Patients
Brief Title: Influence of Thoracic Epidural Anesthesia on Skin Sympathetic Activity and Heart Rate Variability
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Other Study IDs: 01-Anast-04
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2006-03

CONDITIONS: Abdominal Surgery; Abdominothoracic Surgery

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of the study is to evaluate the impact of epidural anesthesia on sympathetic activity in surgical patients. The study investigates whether a segmental sympathetic block can be determined and can be correlated to level of the sensoric blockade.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* combined anesthesia with thoracic epidural anesthesia 8 (Th6-9
* Body-mass-index < 30

Exclusion Criteria:

* Fever, Hypothermia, SIRS
* Microangiopathy
* Neuropathy
* Sensomotoric deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-04; Study Completion 2006-01

PRIMARY OUTCOMES:
Hemodynamic parameters

SECONDARY OUTCOMES:
Level of sensoric block
skin temperature

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Freise, MD, Principal Investigator — Department of Anesthesiology and Intensive Care, University Hospital Münster
Locations (1):
- Department of Anesthesia and Intensive Care, University Hospital Muenster, Münster, Germany

REFERENCES:
- [Result] Freise H, Meissner A, Lauer S, Ellger B, Radke R, Bruewer M, Brodner G, Van Aken HK, Sielenkamper AW, Fischer LG. Thoracic epidural analgesia with low concentration of bupivacaine induces thoracic and lumbar sympathetic block: a randomized, double-blind clinical trial. Anesthesiology. 2008 Dec;109(6):1107-12. doi: 10.1097/ALN.0b013e31818db16c. PMID 19034108